CLINICAL TRIAL: NCT05333653
Title: The Effect of Continous Supportive Care at Childbirth on Maternal Psychological Well-being: A Single-blind Randomized Controlled Trial
Brief Title: Supportive Care During Childbirth and Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gozde Gokce Isbir, Associate Prof, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GIsbir
Record Dates: First submitted 2022-02-02; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Psychological Well-being; Childbirth; Care Pattern, Maternal
Keywords: Intrapartum supportive care; birth trauma; fear of childbirth; maternal attachment; perinatal well-being
MeSH Terms: conditions — Psychological Well-Being; Birth Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continous Supportive Care (Experimental): Participants were provided care in different rooms, blinded to the differences in practice used between the two groups. In the same clinic, a room was designed as a positive delivery room by the researchers and a relaxing environment was created. In this room, supportive care parameters recommended by The Royal College of Midwives (2012) were applied to the women in the ICSC group in line with their preferences.
  Interventions: Other: Continouse supportive care
- Control (Experimental): Participants in the control group, on the other hand, received the routine care given in the hospital by other midwives in the clinic, and there was a change of caregiver midwife during shift changes. The care provided in the hospital during delivery is mostly focused on low level of physical comfort and high level of follow-up.
  Interventions: Other: routine care

INTERVENTIONS:
Other: Continouse supportive care — Participants were provided care in different rooms, blinded to the differences in practice used between the two groups. In the same clinic, a room was designed as a positive delivery room by the researchers and a relaxing environment was created. In this room, supportive care parameters recommended by The Royal College of Midwives (2012) were applied to the women in the ICSC group in line with their preferences.
  Participants in the control group, on the other hand, received routine care given in the hospital by other midwives in the clinic.
  Arms: Continous Supportive Care
Other: routine care — Participants in the control group, on the other hand, received the routine care given in the hospital by other midwives in the clinic, and there was a change of caregiver midwife during shift changes. The care provided in the hospital during delivery is mostly focused on low level of physical comfort and high level of follow-up.
  Arms: Control

SUMMARY:
The aim of this study is to evaluate the effects of continuous supportive care (ICSC) at birth on some parameters of maternal psychological well-being.

DETAILED DESCRIPTION:
This is a single-blind randomized controlled trial. Data were collected from 80 women who gave birth in the obstetrics clinic of a state hospital in the south of Turkey between December 2020 and June 2021. Participants who met the inclusion criteria were informed about the purpose of the study and the procedures to be performed, informed consent was obtained from those who agreed to participate, and women were assigned to the groups in line with a computer-based randomization program with an allocation ratio of 1:1. Block randomization could not be performed because of the different and long delivery processes. Data were collected in both groups at birth (latent phase, active phase, and transitional phase), within 24 hours of birth, and 6th-8th postpartum days after hospital admission and at least one hour of care. collected by the first author. The CONSORT directive was followed in the planning, implementation and writing of the research.

ELIGIBILITY:
Inclusion Criteria:

* The ages of 18-40 women,
* At least primary school graduate,
* Mother tongue Turkish,
* Single fetus,
* Term,
* Spontaneous birth,
* Cervical dilatation between 0-6 cm (latent phase) and without a condition that could prevent vaginal delivery.
* Primiparous and multiparous women
* Not have any disease or complication and agreed to participate in the study were included.

Exclusion Criteria:

* Women who developed a complication with the fetus or themselves during delivery,
* Underwent emergency cesarean section,
* Not be reached during follow-ups by telephone,
* Wanted to withdraw from the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-27 (Actual)

PRIMARY OUTCOMES:
Fear of Childbirth (DFS) | through delivery, an average of 24th hours
  Women's fears at the time of birth were evaluated with the Delivery fear scale (DFS).
  This scale was developed by Wijma et al (2002) for fear during delivery. The Turkish validity and reliability of the scale were performed by Sercekus et al. (2017). This scale consisting of 10 items is a 10-point Likert-type. The positive-meaning items are scored in reverse order. Therefore, the scores ranged from 10 to 100. The scale has no cutoff score, and high scores indicated higher fear.
Perceived control and support in birth (SCIB) | Postpartum 24th hours
  Women's perceptions of support and control at the time of birth were evaluated with the Perceived control and support in birth scale.
  SCIB was developed by Ford et al., (2009) to measure perceived support and control in birth. The Turkish validity and reliability of the scale were performed by Inci et al. (2015). This scale consisting of 33 items is a 5-pointLikert-type (5 = agree completely to 1 = disagree completely). Ten items are scored in reverse order. The scores ranged from 33 to 165. SCIB subscales include internal control, external control, and support. The scale has no cutoff score, higher scores are associated with a higher degree of perceived support and of control during birth. The Cronbach's alpha for the original scale was measured as .95 (Ford et al., 2009) and Turkish version was measured as 0.84 (Inci et al.,2015). In this study, this scale was administered within 24 hours postpartum.
Birth Trauma (City BITS) | Postpartum 8 th week
  Birth trauma of women were evaluated with the City Birth Trauma Scale. City BiTS was developed by Ayers et al., (2018) to measure birth trauma. The Turkish validity and reliability of the scale were performed by Bayrı Bingöl et al. (2021). The scale is a fourpoint Likert-type instrument composed of 29 items. Higher scores reflect greater risk for Post-traumatic Stress Disorder (PTSD). The Cronbach's alpha for the original scale was measured as .92 (Ayers et al.,2018) and Turkish version was measured as 0.91 (Bayrı Bingöl et al., 2021). In this study, 6-8 days after birth to determine whether they meet the criteria for birth trauma and birth-related PTSD.
Maternal Attachment (MAI) | Postpartum 8 th week
  Maternal attachment of women was evaluated with the Maternal Attachment Inventory.
  MAI, was developed by Muller (1994) to measure maternal attachment. The Turkish validity and reliability of the scale were performed by Kavlak et al. (2009). This scale consisting of 26 items is a 4-point Likert-type (4 = every time to 1 = any time). The scores ranged from 26 to 104 and high scores indicated higher maternal attachment. The Cronbach's alpha for the original scale was measured as .76 - .85 at different time (Muller, 1994) and Turkish version was measured as 0.77 (Kavlak et al., 2009). In this study, 6th to 8th postnatal days were used to measure maternal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Gozde Gokce Isbir, Principal Investigator — Mersin University
Locations (1):
- Gozde Gokce Isbir, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No